CLINICAL TRIAL: NCT00824772
Title: Evaluation of Pharmacogenetic Factors Contributing to Dose Requirement of Fentanyl for Postoperative Pain Control: Genetic Polymorphisms of OPRM1, ABCB1, CYP3A4 and CYP3A5
Brief Title: Evaluation of Pharmacogenetic Factors Affecting Fentanyl Requirements for Postoperative Pain Control
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Kye-Min Kim, Associate professor, Department of Anesthesiolgy & Pain Medicine, Inje University, Inje University
Other Study IDs: 00012007317-00
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Pain, Postoperative
Keywords: pharmacogenetics
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Fentanyl is a widely used opioid analgesic. There are big interindividual variabilities in dose requirements of fentanyl for postoperative pain control. This study aims to reveal the genetic factors affecting the variable requirements of fentanyl during postoperative period.

DETAILED DESCRIPTION:
The candidate genes are OPRM1, ABCB1,CYP3A4 and CYP3A5.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total abdominal hysterectomy (TAH) or laparoscopy assisted vaginal hysterectomy (LAVH) under general anesthesia
* Patients who want to use intravenous patient controlled analgesia (PCA) after surgery
* ASA physical status class I, II

Exclusion Criteria:

* history of drug addiction
* opioid medication within 12 hours before surgery
* previous history of opioid medication for 3 months
* neurologic disorder
* cardiac disorder
* hepatic disease
* renal disease
* respiratory disease such as COPD, asthma
* sleep apnea
* BMI > 30
* psycotic disorder

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gynecologic patients undergoing total abdominal hysterectomy or laparoscpy assisted vaginal hysterectomy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kye-Min Kim, MD. PhD., Principal Investigator — Department of Anesthesia, Inje University Sanggye Paik Hospital
Locations (1):
- Inje University Sanggye Paik Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KM, Kim HS, Lim SH, Cheong SH, Choi EJ, Kang H, Choi HR, Jeon JW, Yon JH, Oh M, Shin JG. Effects of genetic polymorphisms of OPRM1, ABCB1, CYP3A4/5 on postoperative fentanyl consumption in Korean gynecologic patients. Int J Clin Pharmacol Ther. 2013 May;51(5):383-92. doi: 10.5414/CP201824. PMID 23557865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Dates of recruitment: 2008 Sep - 2010 Feb
  * Type of location: university hospital
Pre-assignment Details: No group assignment required for this study.
Groups:
- Gynecologic Patients Undergoing TAH, LAVH: * Inclusion criteria:
    19 - 65 years, ASA I,II, total abdominal hysterectomy (TAH) or laparoscopic assisted vaginal hysterectomy (LAVH) under general anesthesia
  * Exclusion criteria history of cardiovascular, renal, hepatic,neurological,psychological, respiratory disease. sleep apnea, or chronic pain or those taking analgesics, obesity
Period: Overall Study
Arm/Group | Gynecologic Patients Undergoing TAH, LAVH
Started | 204
Completed | 196
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Gynecologic Patients Undergoing TAH, LAVH
Number analyzed (Participants) | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 204
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 204

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Cumulative Fentanyl Consumption
Time Frame: 24 hr after surgery
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Gynecologic Patients Undergoing TAH, LAVH
Number analyzed (Participants) | 196
mcg | 836 (416)

2. Secondary Outcome: Postoperative Cumulative Fentanyl Consumption
Time Frame: 48hr after surgery
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Gynecologic Patients Undergoing TAH, LAVH
Number analyzed (Participants) | 196
mcg | 1028 (520)

ADVERSE EVENTS:
Arm/Group | Gynecologic Patients Undergoing TAH, LAVH
Serious Adverse Events (participants affected / at risk) | 0/204
Other Adverse Events (participants affected / at risk) | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No